CLINICAL TRIAL: NCT00385346
Title: Expressive Writing as a Therapeutic Intervention in Male Infertility
Brief Title: Expressive Writing in Male Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Prof. Dr. R. Liedtke, Department of Psychosomatic Medicine and Psychotherapy, University of Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lfd.Nr.068/06
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2009-09

CONDITIONS: Infertility, Male
Keywords: Expressive writing; Male infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- A 1 (Experimental): Expressive writing
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Expressive writing — Patients in the intervention group write on three day for 20 minutes about highly emotional topics In the control group patients write on three days for 20 minutes about topics with relatively low emotional involvement such as diet, time management and sport.

SUMMARY:
The purpose of this study is to determine whether expressive writing can be effective in improving the well-being and sperm quality in patients with male infertility.

DETAILED DESCRIPTION:
Expressive writing is a therapeutic intervention designed by the psychologist James W. Pennebaker. Individuals write on three days for about 20 minutes about particularly stressful experiences in their life. Several studies showed that expressive writing can have beneficial effects on the frequency of health care utilization and well-being. Particularly in patients with rheumatism, kidney cancer and posttraumatic stress disorder expressive writing showed an positive effect on subjective well-being. Furthermore, in several studies expressive writing showed a positive effect on immune parameters.

As many studies suggest an important negative effect of stress on well-being and sperm parameters in male infertility, we want to investigate the effect of expressive writing in male infertility.The expressive writing condition is compared to a non emotional writing condition, in which individuals write about mainly non emotional topics such as time management. In this randomized-controlled trial subjects were allocated sequentially by block wise randomization (block size of 4). For randomization a computer generated random list was used. The allocation was concealed in a series of numbered sealed envelopes. The envelope was opened immediately before the first writing session.

ELIGIBILITY:
Inclusion Criteria:

* Male infertile patients with a pathological spermiogram according to WHO criteria

Exclusion Criteria:

* Drugs affecting sperm quality
* Patients with chromosomal anomalies affecting sperm quality (e.g. Klinefelter- Syndrome)
* Severe Psychiatric disorder defined as psychotic disorder (schizophrenia, bipolar disorder) or substance-related disorder
* Patients currently in psychotherapeutic or psychiatric therapy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Scores on rating scale for perceived stress in infertility | 3 months

SECONDARY OUTCOMES:
Scores on rating scale for personality dimensions | 3 months
Sperm parameters | 3-12 months
Score on rating scale for coping | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Liedtke, MD, Study Chair — University of Bonn, Department of Psychosomatic Medicine
Locations (1):
- University of Bonn, Department of Psychosomatic Medicine, Bonn, Germany

REFERENCES:
- [Background] Smyth J, Helm R. Focused expressive writing as self-help for stress and trauma. J Clin Psychol. 2003 Feb;59(2):227-35. doi: 10.1002/jclp.10144. PMID 12552631
- [Background] de Moor C, Sterner J, Hall M, Warneke C, Gilani Z, Amato R, Cohen L. A pilot study of the effects of expressive writing on psychological and behavioral adjustment in patients enrolled in a Phase II trial of vaccine therapy for metastatic renal cell carcinoma. Health Psychol. 2002 Nov;21(6):615-9. doi: 10.1037//0278-6133.21.6.615. PMID 12433015
- [Background] Petrie KJ, Fontanilla I, Thomas MG, Booth RJ, Pennebaker JW. Effect of written emotional expression on immune function in patients with human immunodeficiency virus infection: a randomized trial. Psychosom Med. 2004 Mar-Apr;66(2):272-5. doi: 10.1097/01.psy.0000116782.49850.d3. PMID 15039514
- [Background] Pennebaker JW. The effects of traumatic disclosure on physical and mental health: the values of writing and talking about upsetting events. Int J Emerg Ment Health. 1999 Winter;1(1):9-18. PMID 11227757
- [Background] Richards JM, Beal WE, Seagal JD, Pennebaker JW. Effects of disclosure of traumatic events on illness behavior among psychiatric prison inmates. J Abnorm Psychol. 2000 Feb;109(1):156-60. doi: 10.1037//0021-843x.109.1.156. PMID 10740948
- [Background] Petrie KJ, Booth RJ, Pennebaker JW. The immunological effects of thought suppression. J Pers Soc Psychol. 1998 Nov;75(5):1264-72. doi: 10.1037//0022-3514.75.5.1264. PMID 9866186
- [Background] Petrie KJ, Booth RJ, Pennebaker JW, Davison KP, Thomas MG. Disclosure of trauma and immune response to a hepatitis B vaccination program. J Consult Clin Psychol. 1995 Oct;63(5):787-92. doi: 10.1037//0022-006x.63.5.787. PMID 7593871
- [Background] Pennebaker JW, Kiecolt-Glaser JK, Glaser R. Disclosure of traumas and immune function: health implications for psychotherapy. J Consult Clin Psychol. 1988 Apr;56(2):239-45. doi: 10.1037//0022-006x.56.2.239. No abstract available. PMID 3372832